CLINICAL TRIAL: NCT02703610
Title: Randomized Trial of Two Analgesics in Elderly ED Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants were enrolled and the study will not be conducted.
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Andrew Chang, Professor, Albany Medical College
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 4733
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pain
Keywords: Pain; Elderly
MeSH Terms: conditions — Pain | interventions — oxycodone-acetaminophen; Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycodone/acetaminophen (Active Comparator): Oxycodone/acetaminophen (5 mg/325 mg)
  Interventions: Drug: Oxycodone/acetaminophen
- Ibuprofen/acetaminophen (Active Comparator): Ibuprofen/acetaminophen (400 mg/500 mg)
  Interventions: Drug: Ibuprofen/acetaminophen

INTERVENTIONS:
Drug: Oxycodone/acetaminophen — Patients will be discharged home with a 3 day supply of oxycodone/acetaminophen
  Other Names: Percocet
  Arms: Oxycodone/acetaminophen
Drug: Ibuprofen/acetaminophen — Patients will be discharged home with a 3 day supply of ibuprofen/acetaminophen
  Arms: Ibuprofen/acetaminophen

SUMMARY:
The purpose of this study is to perform a randomized, double blind 2-arm clinical trial of the comparative efficacy of 2 oral analgesics in the the management of acute pain in elderly patients who present and then are discharged from the ED.

DETAILED DESCRIPTION:
To perform a randomized, double blind 2-arm clinical trial of the comparative efficacy of 2 oral analgesics in the the management of acute pain in elderly patients who present and then are discharged from the ED.. The 2 groups are as follows:

1. Oxycodone/acetaminophen (5/325)
2. Ibuprofen/acetaminophen (400/500)

ELIGIBILITY:
Inclusion Criteria:

* Complaint of acute pain of < 7 days duration
* ED attending plans to discharge patient home with an oral analgesic

Exclusion Criteria:

* Inability to confirm reliable means of phone followup.
* Past use of methadone
* Chronic condition requiring frequent pain management such as sickle cell disease, fibromyalgia, or any neuropathy
* History of an adverse reaction to any of the study medications
* Ibuprofen or acetaminophen or opioids taken in past 4 hours
* History of peptic ulcer disease
* Report of any prior use of recreational narcotics
* Medical condition that might affect metabolism of opioid analgesics, acetaminophen, or ibuprofen such as hepatitis, renal insufficiency, hypo- or hyperthyroidism, Addison's or Cushing's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Between group difference in change in NRS pain scores | 24 hours
  Between group difference in change in NRS pain scores at 24 hours

SECONDARY OUTCOMES:
Between group difference in change in NRS pain scores at first followup contact | 24-72 hours
  Between group difference in change in NRS pain scores at first followup contact
Between group difference in change in NRS pain scores | 48 hours and 72 hours
  Between group difference in change in NRS pain scores at 48 hours and 72 hours
Between group difference in side effects | 24 hours, 48 hours and 72 hours
  Proportion with side effects (nausea, vomiting, pruritus, dizziness, drowsiness, constipation)
Change in NRS pre and 2 hours post most recent dose of pain medication taken | 24 hours
  Change in NRS pre and 2 hours post most recent dose of pain medication taken
Between group difference in Likert pain scores | 24, 48, and 72 hours
  Pain evaluation on a 4 point Likert scale (none, mild, moderate, severe)
Satisfaction | 24, 48, and 72 hours
  Satisfaction assessed by 4-point Likert Scale: very satisfied, satisfied, unsatisfied, very unsatisfied
Between group differences in NRS pain scores in patients who have extremity injuries, extremity fractures, and 10/10 pain. | 24-72 hours
  Between group differences in NRS pain scores in patients who have extremity injuries, extremity fractures, and 10/10 pain.
Difference in percentage of physicians and patients in each group who successfully identified which study group the patient had been randomized to | 24-72 hours
  Difference in percentage of physicians and patients in each group who successfully identified which study group the patient had been randomized to
Want same medication again | 24-72 hours
  Between group difference in proportion of patients who would want the same medication again

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No